CLINICAL TRIAL: NCT03027206
Title: Effects of Vibration Techniques and Expiratory Flow Acceleration in Premature Pain Parameters With Pneumonia
Brief Title: Respiratory Physiotherapy Change Premature Pain With Pneumonia
Acronym: RPCPPWP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Amazon University (Other)
Collaborators: Fundação Santa Casa de Misericórdia do Pará (FSCMPA) (Unknown)
Responsible Party: Principal Investigator, Paulo Eduardo Santos Avila, Assistant teacher, Amazon University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1.690.842
Record Dates: First submitted 2016-11-21; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Premature; Pneumonia; Pain; Physiotherapy
MeSH Terms: conditions — Premature Birth; Pneumonia; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vibration technique (Experimental): Rhythmic and rapid movements of isometric contraction of the forearm, applied manually over the anterior region of the thorax
  Interventions: Other: Vibration technique
- Acceleration of expiratory flow (Experimental): Soft compression of the thorax applied with one hand on the lower ribs and the other using the ulnar border on the supramammary line
  Interventions: Other: Acceleration of expiratory flow

INTERVENTIONS:
Other: Vibration technique — Comparison of different technique
  Arms: Vibration technique
Other: Acceleration of expiratory flow — Comparison of different technique
  Arms: Acceleration of expiratory flow

SUMMARY:
Objective to evaluate the effects of vibration techniques and acceleration of expiratory flow on pain parameters in preterm infants diagnosed with pneumonia hospitalized in the Intensive Care Unit and Neonatal Intermediate Care Unit. The Method is a descriptive and interventional study, in which 28 PTNB were randomly divided into two groups: Group 1 submitted to the vibration technique and Group 2 - to the acceleration of the expiratory flow, both techniques were applied in an interval of up to ten minutes, for Three consecutive days. The pain indicators were evaluated according to the PIPP scale in three moments. For statistical analysis, the Friedman tests and Variance Analysis were applied, the level of significance adopted was 5%.

DETAILED DESCRIPTION:
A descriptive, longitudinal, quantitative approach was carried out in which 28 preterm infants with diagnosis of pneumonia hospitalized in the NICU and NICU of the Santa Casa de Misericórdia Foundation of Pará (FSCMPA) participated in the study period from July to October 2016. The research obeyed ethical principles Of Resolution 466/12 of the National Health Council (CNS) and was initiated after approval by the Research Ethics Committee of the FSCMPA, opinion 1,690,842. The selection criteria were obtained through the collection of data from the records of newborns and annotated in standardized charts. Once included in the study, the patients were randomly divided into two groups of 14 PTNB, the premature group 1 were submitted to the vibration technique (rhythmic and rapid movements of isometric contraction of the forearm, applied manually over the anterior chest region) and the Of Group 2 to the acceleration of the expiratory flow (soft compression of the thorax applied with one hand in the lower ribs and the other using the ulnar border on the supramammary line). Both techniques were performed with the premature dorsal position, at the time of the expiratory phase, with a maximum duration of 10 minutes, once a day, for three consecutive days, in the afternoon period and by the same physiotherapist. After this procedure, aspiration of the upper airways of premature infants was performed. The pain indicators of the preterm infants (PIPP) of the two groups were evaluated in three moments, before the application of the technique (T1), immediately after the application of the technique (T2) and 15 minutes After its completion (T3), by a researcher previously trained and blind regarding the procedure performed. PIPP is a multidimensional instrument that evaluates pain indicators in the newborn using the following parameters: gestational age and alertness (contextual factors), heart rate and peripheral oxygen saturation (physiological indicators) that were measured by means of a pulse oximeter Of the brand (Dixtal®) and three aspects of facial mimetics (behavioral factors). Their scores may range from 0 to 21, scores less than or equal to 6 indicate absence of pain, scores above 6 represent mild pain and scores higher than 12 indicate the presence of moderate to severe pain.

ELIGIBILITY:
Inclusion Criteria:

* Included in this study were RNPT of both genders, of low weight (1500 to 2500g) or normal weight (over 2500g).
* With clinical diagnosis of pneumonia.
* Who were on spontaneous ventilation (ambient air or with the aid of oxygen therapy).
* Agreed to participate in the research, through the signing of the Informed Consent Form for minors.

Exclusion Criteria:

* Newborns with a gestational age greater than 37 weeks.
* With diseases or procedures that cause pain in the newborn such as necrotizing enterocolitis, thoracotraumatis, thoracic or abdominal drainage, and umbilical catheter.
* Who were less than 72 hours Life with birth weight less than 1500g (very low weight and extreme low weight).
* As well as those who underwent invasive or non-invasive mechanical ventilation.
* Sedated.
* With vasoactive drugs or medications that interfered in the physiological parameters of pain.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of the parameters of the pain profile scale in preterm infants at different times | The total collection period was six months, and each procedure was performed on the volunteers for three consecutive days.
  The pain indicators of the preterm infants (PIPP) of the two groups were evaluated in three moments, before the application of the technique (T1), immediately after the application of the technique (T2) and 15 minutes After its termination (T3), by a researcher previously trained and blind as to the procedure performed

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Patel RM, Kandefer S, Walsh MC, Bell EF, Carlo WA, Laptook AR, Sanchez PJ, Shankaran S, Van Meurs KP, Ball MB, Hale EC, Newman NS, Das A, Higgins RD, Stoll BJ; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Causes and timing of death in extremely premature infants from 2000 through 2011. N Engl J Med. 2015 Jan 22;372(4):331-40. doi: 10.1056/NEJMoa1403489. PMID 25607427
- [Result] Walker CLF, Rudan I, Liu L, Nair H, Theodoratou E, Bhutta ZA, O'Brien KL, Campbell H, Black RE. Global burden of childhood pneumonia and diarrhoea. Lancet. 2013 Apr 20;381(9875):1405-1416. doi: 10.1016/S0140-6736(13)60222-6. Epub 2013 Apr 12. PMID 23582727
- [Result] Brandao AM, Domingues AP, Fonseca EM, Miranda TM, Belo A, Moura JP. [Premature labour with or without preterm premature rupture of membranes: maternal, obstetric and neonatal features]. Rev Bras Ginecol Obstet. 2015 Sep;37(9):428-33. doi: 10.1590/SO100-720320150005283. Portuguese. PMID 26352946
- [Result] Stevens B, Yamada J, Ohlsson A, Haliburton S, Shorkey A. Sucrose for analgesia in newborn infants undergoing painful procedures. Cochrane Database Syst Rev. 2016 Jul 16;7(7):CD001069. doi: 10.1002/14651858.CD001069.pub5. PMID 27420164
- [Result] Als H, Duffy FH, McAnulty GB, Rivkin MJ, Vajapeyam S, Mulkern RV, Warfield SK, Huppi PS, Butler SC, Conneman N, Fischer C, Eichenwald EC. Early experience alters brain function and structure. Pediatrics. 2004 Apr;113(4):846-57. doi: 10.1542/peds.113.4.846. PMID 15060237
- [Result] Silva YP, Gomez RS, Maximo TA, Silva AC. [Pain evaluation in neonatology.]. Rev Bras Anestesiol. 2007 Oct;57(5):565-74. Portuguese. PMID 19462133